CLINICAL TRIAL: NCT06821997
Title: A Phase 2 Clinical Trial of Nalirifox as Neoadjuvant Treatment for Patients With Borderline Resectable Pancreatic Ductal Adenocarcinoma (Nectar Study)
Brief Title: NALIRIFOX Before Surgery for the Treatment of Borderline Resectable Pancreatic Ductal Adenocarcinoma, Nectar Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-4064824; NCI-2025-00732 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-4064824 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Borderline Resectable Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Specimen Handling; Fluorouracil; dehydroftorafur; irinotecan sucrosofate; Leucovorin; Oxaliplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (NALIRIFOX) (Experimental): Patients receive liposomal irinotecan IV over 90 minutes, oxaliplatin IV over 120 minutes, leucovorin IV over 30 minutes and fluorouracil IV over 48 hours on day 1 of each cycle. Cycles repeat every 14 days for 4-8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo surgical resection 4-8 weeks after the last treatment dose. Starting 4-12 weeks after surgery, patients receive liposomal irinotecan, oxaliplatin, leucovorin, and fluorouracil for up to 4 additional cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Irinotecan Sucrosofate; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Irinotecan Sucrosofate — Given IV
  Other Names: inotecan Hydrochloride as Sucrosulfate Salt Form Liposomal Formulation; Irinotecan Liposome; Irinotecan Sucrosofate Liposome; Irinotecan Sucrosofate-containing Pegylated Liposomal Formulation; MM 398; MM-398; MM398; nal-IRI; Nanoliposomal Irinotecan; Nanoliposomal Irinotecan as Sucrosofate; Nanoparticle Liposome Formulation of Irinotecan; Onivyde; PEP 02; PEP-02; PEP02
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
Procedure: Surgical Procedure — Undergo surgical resection
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase II trial tests how well liposomal irinotecan, oxaliplatin, 5-fluorouracil and leucovorin (NALIRIFOX) before surgery works in treating patients with pancreatic ductal adenocarcinoma that is close to major blood vessels, but is still potentially removable by surgery (borderline resectable). Irinotecan is in a class of antineoplastic medications called topoisomerase I inhibitors. It blocks a certain enzyme needed for cell division and deoxyribonucleic acid (DNA) repair and may kill tumor cells. Liposomal irinotecan is a form of the anticancer drug irinotecan that is contained inside very tiny, fat-like particles. Liposomal irinotecan may have fewer side effects and work better than other forms of the drug. Oxaliplatin is in a class of medications called platinum-containing antineoplastic agents. It damages the cell's DNA and may kill tumor cells. 5-fluorouracil, a type of antimetabolite, stops cells from making DNA and it may kill tumor cells. Leucovorin, a form of folic acid, is used to lessen the toxic effects of substances that block the action of folic acid. It is a type of chemoprotective agent and a type of chemosensitizing agent. Giving NALIRIFOX before surgery may improve the chance of successful surgery and decrease the chance of the cancer returning after surgery in patients with borderline resectable pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the antitumor efficacy of the combination of irinotecan sucrosofate (liposomal irinotecan), oxaliplatin and infusional fluorouracil (5-fluorouracil)/leucovorin calcium (leucovorin) (NALIRIFOX) in patients with borderline resectable pancreatic ductal adenocarcinoma.

SECONDARY OBJECTIVES:

I. To evaluate clinical efficacy and tolerability of the proposed treatment regimen.

II. To determine the safety of liposomal irinotecan, oxaliplatin and infusional fluorouracil in patients with borderline resectable pancreatic ductal adenocarcinoma.

EXPLORATORY OBJECTIVES:

I. To evaluate blood-based biomarkers predictive of short- and long-term outcomes.

II. To generate tumor tissue-based biomarkers predictive of short- and long-term outcomes.

OUTLINE:

Patients receive liposomal irinotecan intravenously (IV) over 90 minutes, oxaliplatin IV over 120 minutes, leucovorin IV over 30 minutes and fluorouracil IV over 48 hours on day 1 of each cycle. Cycles repeat every 14 days for 4-8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo surgical resection 4-8 weeks after the last treatment dose. Starting 4-12 weeks after surgery, patients receive liposomal irinotecan, oxaliplatin, leucovorin, and fluorouracil for up to 4 additional cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) and blood sample collection throughout the study.

After completion of study treatment, patients are followed up within 30 days, every 3-6 months for 2 years, then every 6-12 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Have histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC) that is borderline resectable (BR) using the National Comprehensive Cancer Network criteria
* Have a documented Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Absolute neutrophil count (ANC) ≥ 1,500 cells/uL without the use of hematopoietic growth factors
* Platelet count ≥ 100,000 cells/uL
* Hemoglobin ≥ 9 g/dL
* Plasma total bilirubin ≤ upper limit of normal (ULN) (biliary drainage is allowed for biliary obstruction)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Creatine clearance of > 30 mL/min (per Cockroft-Gault equation)
* Plasma albumin ≥ 3 g/dL
* Have measurable or evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an independent ethics committee/institutional review board approved written informed consent form (ICF) prior to receiving any study related procedure

Exclusion Criteria:

* Patients who have had previous chemotherapy or radiotherapy for PDAC
* Patients with resectable, unresectable, or metastatic PDAC
* Presence of germline glucuronosyltransferase (UGT) 1A1 (*28 or *6) or dihydropyrimidine dehydrogenase (DPD) polymorphisms (DPYD*2A [rs3918290, c.1905+1G>A, IVS14+1G>A], c.2846A>T [rs67376798, D949V], c.1679T>G [rs55886062, DPYD*13, I560S], and c.1236G>A [rs56038477, E412E, in haplotype B3]) known to significantly impact CPT-11 and fluorouracil metabolism and associated with increased risk for toxicities
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | Up to 5 years
  MPR will be defined as either complete pathologic response or minimal residual cancer based on the American College of Pathology system. The MPR status will be summarized using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 5 years
  Will be assessed using Response Evaluation Criteria in Solid Tumors 1.1. ORR will be summarized using frequencies and relative frequencies. Estimates of rates will be obtained with 90% credible regions obtained by Jeffrey's prior method.
CA19-9 response rate | Up to 5 years
  Will be summarized using frequencies and relative frequencies. Estimates of rates will be obtained with 90% credible regions obtained by Jeffrey's prior method.
Carcinoembryonic antigen response rate | Up to 5 years
  Will be summarized using frequencies and relative frequencies. Estimates of rates will be obtained with 90% credible regions obtained by Jeffrey's prior method
Positive margin resection rate | Up to 5 years
  Will be summarized using frequencies and relative frequencies. Estimates of rates will be obtained with 90% credible regions obtained by Jeffrey's prior method
Disease-free survival | From start of neoadjuvant therapy until disease progression, subsequent therapy, death due to any cause, or last follow-up, assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods, where estimates of the median times will be obtained with 90% confidence intervals.
Overall survival | From start of neoadjuvant therapy until death due to any cause, or last follow-up, assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods, where estimates of the median times will be obtained with 90% confidence intervals
Incidence of adverse events | Up to 30 days after the last intervention, or until the event has resolved, the study participant is lost to follow-up, the start of a new treatment, or until the study investigator assesses the event(s) as stable or irreversible
  Will be described and graded using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Will be summarized by attribution and grade using frequencies and relative frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Fountzilas, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States